CLINICAL TRIAL: NCT05753670
Title: Effect of Preoperative Single-dose Tamsulosin on Postoperative Urinary Retention After Mid-urethral Sling Placement: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Preoperative Tamsulosin on Postoperative Urinary Retention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Ghazaleh Rostami Nia, Director of Research Division of Urogynecology, NorthShore University HealthSystem, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EH22-470
Record Dates: First submitted 2022-12-13; First posted 2023-03-03 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Retention of Urine
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized, double-blinded, placebo- controlled trial of patients who are undergoing elective mid-urethral sling placement with the Center for Pelvic Health at the Northshore University Health System. Written consent will be obtained.
  Patients who are undergoing a mid-urethral sling placement will be enrolled (after an informed consent discussion) to receive either a single tablet of tamsulosin 0.4mg or a placebo in the preoperative holding area on the day of their scheduled surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will occur by simple randomization with a computer-generated random number list. The patient will be randomized to one of the two groups (preoperative tamsulosin 0.4mg tablet versus placebo). This random number list will be sent directly from the statistician to the pharmacy. The clinician will place an order for the preoperative trial medication and the pharmacy will dispense either a single tablet of tamsulosin 0.4mg or placebo to the preoperative holding area according to the randomization list that the pharmacy has been provided by the statistician. The trial medication will be sent from the pharmacy to the preoperative area to be taken prior to surgery. The clinicians, preoperative and postoperative nursing staff, and the patients will be blinded to the trial group and medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tamsulosin (Experimental): Subjects randomized to the experimental arm will receive a single dose of 0.4mg Tamsulosin tablet in the preoperative holding area prior to their scheduled mid-urethral sling placement in the operating room.
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator): Subjects randomized to the control arm will receive a single dose of a placebo tablet in the preoperative holding area prior to their scheduled mid-urethral sling placement in the operating room.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Subjects randomized to the experimental arm will receive a single dose of 0.4mg Tamsulosin tablet in the preoperative holding area prior to their scheduled mid-urethral sling placement in the operating room.
  Arms: Tamsulosin
Drug: Placebo — Subjects randomized to the control arm will receive a single dose of a placebo tablet in the preoperative holding area prior to their scheduled mid-urethral sling placement in the operating room.
  Arms: Placebo

SUMMARY:
Approximately 25-30% of patients experience postoperative urinary retention after female pelvic surgery with mid-urethral sling placement. These patients are discharged home with a foley catheter for a few days. Despite being common, many patients consider being discharged home with a foley catheter as a complication of surgery and as the worst part of their experience. Previous studies have demonstrated that 3-5 days of preoperative tamsulosin (a safe and low-cost medication) have been shown to improve postoperative urinary retention rates. Although it takes tamsulosin 5 days to reach a steady-state in a patient, it reaches peak blood volume in 4-5 hours in a fasting patient. The effect of a single dose of preoperative tamsulosin on postoperative urinary retention has not been studied, however would be substantially easier for patients than multiple days of preoperative doses. In this study, the investigators would like to give patients preoperative tamsulosin versus placebo. The investigators would then evaluate for postoperative urinary retention. Previous studies have demonstrated a postoperative urinary retention rate decrease of 65-88% after various tamsulosin protocols. However, the effect of single preoperative dose of tamusloin on postoperative urinary retention has yet to be studied in female pelvic surgery. The investigators hypothesize that a single preoperative dose of tamsulosin will decrease the number of patients with postoperative urinary retention and therefore discharged with a foley catheter. Our goal is to improve patient outcomes and satisfaction postoperatively.

DETAILED DESCRIPTION:
Postoperative urinary retention has been defined as the inability to void despite having fluid in the bladder during the postoperative period. Urinary retention after pelvic reconstructive surgery requiring indwelling catheter or self-catheterization usage occurs in approximately 30-60% of patients postoperatively.

During a retro-fill voiding trial, the bladder is back-filled with a set amount of sterile water (often 300mL), the catheter is removed, the patient is permitted to void and the voided volume is compared with a bladder scan post void residual volume. "Passing" a voiding trial has previously been defined as voiding equal or greater than ⅔ the residual volume, whereas others characterize "passing" as voiding at least 200mL and voiding a greater volume than the post-void residual volume. If the patient does not "pass" the voiding trial, the patient is characterized as having postoperative urinary retention and is discharged home with an indwelling catheter to prevent detrusor injury from bladder over-distention, pain and urinary tract infection.

Many women consider being discharged home with a foley catheter to be a surgical complication and describe catheter use as the worst aspect of their surgery. Indwelling catheters are the leading cause of hospital-acquired urinary tract infections (UTIs), are often a source of embarrassment and inconvenience for patients, and often require additional office visits and healthcare utilization.

Tamsulosin is an alpha-adrenergic receptor blocker which is thought to increase smooth muscle relaxation and improve urinary flow. Current literature has been primarily focused on the effect of tamsulosin in men with benign prostatic hyperplasia, however may be beneficial in women as well with limited studies for postoperative urinary retention. Chapman, et al published a randomized control trial evaluating postoperative urinary retention after female pelvic reconstructive surgery. These patients underwent 10 days of tamsulosin (3 days preoperative and 7 days postoperative) and were found to have a 65% decrease in the urinary retention rate from 25.8% to 8.8%. Livne, et al published a study evaluating postoperative urinary retention decrease of 79.2% after postoperative administration of dibenzyline (an alpha-adrenergic receptor blocker) in women undergoing hysterectomy (post-operative urinary retention rate of 18.75% in controls and 3.9% in the treatment group). Additional studies have also been published evaluating postoperative urinary retention in men and women undergoing various surgeries and have demonstrated a decrease in postoperative urinary retention after tamsulosin administration from 72-88% compared with controls. These studies vary in tamsulosin administration from multiple days preoperative and postoperative to multiple doses preoperative and postoperative to a single postoperative dose, however no studies have been published in evaluating a single preoperative dose of tamsulosin and the effect on postoperative urinary retention. This has previously been studied as tamsulosin reaches a steady state in approximately 5 days, however when tamsulosin is given in a fasting patient, it can reach the maximum blood concentration in approximately 4-5 hours. As the majority of female pelvic reconstructive surgeries performed by our department are same-day surgeries, with patients being discharged the day of surgery, the investigators would like to investigate the effect of a single preoperative dose of tamsulosin on postoperative urinary retention and, by effect, home catheter usage after surgery. Tamsulosin is cost-effective at approximately $2 per tablet. Despite primarily being prescribed for benign prostatic hyperplasia, tamsulosin has been found to be a safe and well-tolerated treatment for voiding dysfunction in women.

Postoperative urinary retention is common after pelvic reconstructive surgery with mid-urethral sling placement and is extremely bothersome to patients. Tamsulosin is a low-risk, well tolerated, cost-effective medication that studies have suggested may decrease the rate of postoperative urinary retention. No study to date has evaluated preoperative administration of single- dose tamsulosin for postoperative urinary retention in a randomized placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Mid-urethral sling placement

Exclusion Criteria:

* Age <18
* Planned combined cases with colorectal surgery, general surgery, or gynecology-oncology
* Planned sling revision or history of prior sling placement
* Known history of urinary retention
* Concomitant intravesical botulinum injections
* Known contraindication to tamsulosin

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-06-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University Health System, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willis-Gray MG, Wu JM, Field C, Pulliam S, Husk KE, Brueseke TJ, Geller EJ, Connolly A, Dieter AA. Is a Postvoid Residual Necessary? A Randomized Trial of Two Postoperative Voiding Protocols. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e256-e260. doi: 10.1097/SPV.0000000000000743. PMID 31157716
- [Background] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Background] Wang R, Won S, Haviland MJ, Von Bargen E, Hacker MR, Li J, Lefevre R. Voiding trial outcome following pelvic floor repair without incontinence procedures. Int Urogynecol J. 2016 Aug;27(8):1215-20. doi: 10.1007/s00192-016-2975-y. Epub 2016 Feb 17. PMID 26886553
- [Background] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Background] Pomajzl AJ, Siref LE. Postoperative Urinary Retention. 2023 Jul 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK549844/ PMID 31751034
- [Background] Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003 Dec;189(6):1551-7; discussion 1557-8. doi: 10.1016/s0002-9378(03)00932-3. PMID 14710061
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Propst K, Tunitsky-Bitton E, O'Sullivan DM, Steinberg AC, LaSala C. Phenazopyridine for Evaluation of Ureteral Patency: A Randomized Controlled Trial. Obstet Gynecol. 2016 Aug;128(2):348-355. doi: 10.1097/AOG.0000000000001472. PMID 27399998
- [Background] Meyer LE, Brown JN. Tamsulosin for voiding dysfunction in women. Int Urol Nephrol. 2012 Dec;44(6):1649-56. doi: 10.1007/s11255-012-0275-0. Epub 2012 Sep 16. PMID 22983886
- [Background] Chapman GC, Sheyn D, Slopnick EA, Roberts K, El-Nashar SA, Henderson JW, Mangel J, Hijaz AK, Pollard RR, Mahajan ST. Tamsulosin vs placebo to prevent postoperative urinary retention following female pelvic reconstructive surgery: a multicenter randomized controlled trial. Am J Obstet Gynecol. 2021 Sep;225(3):274.e1-274.e11. doi: 10.1016/j.ajog.2021.04.236. Epub 2021 Apr 21. PMID 33894146
- [Background] Livne PM, Kaplan B, Ovadia Y, Servadio C. Prevention of post-hysterectomy urinary retention by alpha-adrenergic blocker. Acta Obstet Gynecol Scand. 1983;62(4):337-40. doi: 10.3109/00016348309156234. PMID 6138916
- [Background] Madani AH, Aval HB, Mokhtari G, Nasseh H, Esmaeili S, Shakiba M, Shakiba RS, Seyed Damavand SM. Effectiveness of tamsulosin in prevention of post-operative urinary retention: a randomized double-blind placebo-controlled study. Int Braz J Urol. 2014 Jan-Feb;40(1):30-6. doi: 10.1590/S1677-5538.IBJU.2014.01.05. PMID 24642148
- [Background] Chapman GC, Sheyn D, Petrikovets A, Mahajan ST, El-Nashar S, Pollard R, Mangel JM. Tamsulosin to Prevent Postoperative Urinary Retention After Female Pelvic Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2020 Nov;26(11):682-687. doi: 10.1097/SPV.0000000000000650. PMID 30418263
- [Background] Mohammadi-Fallah M, Hamedanchi S, Tayyebi-Azar A. Preventive effect of tamsulosin on postoperative urinary retention. Korean J Urol. 2012 Jun;53(6):419-23. doi: 10.4111/kju.2012.53.6.419. Epub 2012 Jun 19. PMID 22741052
- [Background] Wilde MI, McTavish D. Tamsulosin. A review of its pharmacological properties and therapeutic potential in the management of symptomatic benign prostatic hyperplasia. Drugs. 1996 Dec;52(6):883-98. doi: 10.2165/00003495-199652060-00012. PMID 8957159
- [Background] Buckley BS, Sanders CD, Spineli L, Deng Q, Kwong JS. Conservative interventions for treating functional daytime urinary incontinence in children. Cochrane Database Syst Rev. 2019 Sep 18;9(9):CD012367. doi: 10.1002/14651858.CD012367.pub2. PMID 31532563

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Tamsulosin
Started | 90 | 89
Completed | 81 | 80
Not Completed | 9 | 9
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin | Placebo | Total
Number analyzed (Participants) | 80 | 81 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (2) | 56.4 (2) | 56.5 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 81 | 161
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 26
  Not Hispanic or Latino | 65 | 70 | 135
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 63 | 56 | 119
  More than one race | 12 | 16 | 28
  Unknown or Not Reported | 0 | 2 | 2
Current smoker [Count of Participants; unit: Participants] | 3 | 6 | 9
Postmenopausal [Count of Participants; unit: Participants] | 49 | 45 | 94
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.88 (5.97) | 27.82 (5.42) | 28.35 (5.71)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Urinary Retention
Description: Determine the postoperative urinary retention rates after preoperative administration of tamsulosin compared with placebo. This will be determined immediately postoperative in the postoperative recovery room based on whether patients pass or fail their voiding trial described above. The result will be documented in electronic medical records and obtained from chart review.
Time Frame: Immediate postoperative evaluation (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 80 | 81
Participants | 14 | 16

2. Secondary Outcome: Number of Participants With Postoperative Urinary Tract Infection (UTI)
Description: Compare differences in the incidence of postoperative UTI (number of participants diagnosed with a UTI within 30 days of procedure) after preoperative administration of tamsulosin compared with placebo.
Time Frame: Chart review of 30 days postoperative after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 80 | 81
Participants | 1 | 1

3. Secondary Outcome: Number of Participants With Unplanned Admission or Unplanned Healthcare Encounter
Description: Evaluate the difference in unplanned admission the day or surgery or unplanned admission within 30 days after surgery, unplanned office visits within 30 days after surgery or Northshore encounters within 30 days after surgery after preoperative administration tamsulosin compared with placebo. These medical encounters will include any need for additional medical treatment, phone calls, complications or patient concerns within 30 days postoperatively. This data will be collected via chart review.
Time Frame: Chart review of 30 days postoperative after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 80 | 81
Participants | 6 | 4

4. Secondary Outcome: Number of Participants With Postoperative Hypotension or Syncope
Description: Compare the number of participants with hypotension or syncope (immediately postoperative) after preoperative administration of tamsulosin compared with placebo.
Time Frame: Immediate postoperative evaluation (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 80 | 81
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Tamsulosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/81
Other Adverse Events (participants affected / at risk) | 0/80 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05753670/Prot_SAP_000.pdf